CLINICAL TRIAL: NCT02035241
Title: Investigation on Effect of Herbs and Spices on Glucose and Insulin Responses, Anti-inflammatory Properties, Antioxidative Capacity and Satiety in Healthy Subjects
Brief Title: Effect of Herbs and Spices on Metabolic Regulation and Appetite in Healthy Subjects
Acronym: AFC-SPICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Elin Östman, Assoc. Prof, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LUND-AFC-STAGE3-SPICES
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Spices; Herbs; Functional food; Cardiometabolic risk; Metabolic syndrome; Inflammation; Appetite; Gut hormone
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Spices 1 (Experimental): 220 ml test drink containing spices 1, acute study / one time administration
  Interventions: Dietary Supplement: Spices 1
- Spices 2 (Experimental): 220 ml test drink containing spices 2, acute study / one time administration
  Interventions: Dietary Supplement: Spices 2
- Spices 3 (Experimental): 220 ml test drink containing spices 3, acute study / one time administration
  Interventions: Dietary Supplement: Spices 3
- Herbs 1 (Experimental): 220 ml test drink containing herbs 1, acute study / one time administration
  Interventions: Dietary Supplement: Herbs 1
- Herbs 2 (Experimental): 220 ml test drink containing herbs 2, acute study / one time administration
  Interventions: Dietary Supplement: Herbs 2
- Placebo (Placebo Comparator): 220 ml control drink, acute study / one time administration
  Interventions: Dietary Supplement: Control drink

INTERVENTIONS:
Dietary Supplement: Spices 1 — In this study, subjects are asked to consume 200 ml beverage drinks contain certain amounts of spices 1. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Spices 1
Dietary Supplement: Spices 2 — In this study, subjects are asked to consume 200 ml beverage drinks contain certain amounts of spices 2. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Spices 2
Dietary Supplement: Spices 3 — In this study, subjects are asked to consume 200 ml beverage drinks contain certain amounts of spices 3. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Spices 3
Dietary Supplement: Herbs 1 — In this study, subjects are asked to consume 200 ml beverage drinks contain certain amounts of herbs 1. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Herbs 1
Dietary Supplement: Herbs 2 — In this study, subjects are asked to consume 200 ml beverage drinks contain certain amounts of herbs 2. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Herbs 2
Dietary Supplement: Control drink — As a control, subjects are asked to consume 200 ml control drinks. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate how herbs and spices affect acute/postprandial glucose and insulin responses, inflammatory markers, appetite control peptides, antioxidative capacity, as well as subjective appetite ratings (VAS-visual analogue scales) in healthy volunteers. We hypothesize that certain herbs and spices added to a standardized meal will improve postprandial glucose tolerance and other metabolic biomarkers in healthy volunteers, compared with a similar meal without the corresponding plant materials.

DETAILED DESCRIPTION:
The aims of the study is to investigate whether consumption of preload isovolumetric (220 ml) spice-based beverages contained total polyphenol concentration to 185 mg gallic-acid equivalents followed by white wheat bread challenge (contained 50 g available carbohydrate) might affect postprandial glucose metabolism, inflammatory markers, appetite-related gut hormones, plasma antioxidant capacity, as well as appetite sensations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Signed informed consent
* BMI 20 - 28 kg/m2 with weight change <3 kg latest 2 months)
* Must be able to accept herbs and spices

Exclusion Criteria:

* Below 18 years
* Uncomfortable speaking English and/or difficulties in understanding spoken English
* Smoking or using snuff
* Vegetarian or vegan
* Stressed by venous blood sampling or previous experience of being difficult to cannulate
* Receiving any drug treatment that may influence the study outcomes
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changing on blood glucose concentration after treatment with herbs and spices | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  The capillary blood samples will be taken for blood glucose analysis

SECONDARY OUTCOMES:
Changing on subjective appetite ratings after treatment with herbs and spices | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  Appetite will be assessed using standard subjective 100 mm VAS (visual analogue scale) at time intervals throughout each visit
Changing on metabolic biomarkers after treatment with herbs and spices | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  The venous blood samples will be taken for insulin, inflammatory markers (i.e. interleukin-6, interleukin-8, tumor necrosis factor-alpha, necrosis factor kappa-beta, adiponectin and C-reactive protein), appetite-related gut hormones (i.e. glucagon-like peptide-1 and peptide tyrosine-tyrosine)
Changing on urine metabolite profile after treatment with herbs and spices | Prior to the initial intervention at 0 min and up to 24-h after intervention
  Metabolite profile will be analyzed using Liquid Chromatography-Mass Spectrometry based methods
Changing on plasma metabolite profile after treatment with herbs and spices | Prior to the initial intervention at 0 min and after intervention at 60, 90, 120, 180 min.
  Metabolite profile will be analyzed using Liquid Chromatography-Mass Spectrometry based methods

CONTACTS AND LOCATIONS:
Overall Officials: Elin Östman, PhD, Principal Investigator — Lund University; Yoghatama Cindya Zanzer, MSc, Principal Investigator — Lund University
Locations (1):
- Antidiabetic Food Centre (Medicon Village) - Lund University, Lund, Skåne County, Sweden

REFERENCES:
- See also: Antidiabetic Food Centre - Vinnova Excellence Centre in Research and Innovation at Lund University, SWEDEN — http://portal.research.lu.se/portal/sv/projects/antidiabetic-food-centre(3a9bae87-b64a-49f5-97a4-868a8bb776ae).html